CLINICAL TRIAL: NCT01804608
Title: Kinematics of Lower Limb, Pain and Function of the Women With Patellofemoral Pain Syndrome Who Underwent Two Types Treatment: Randomized Clinical Trial
Brief Title: Kinematics of Lower Limb, Pain and Function of the Women With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Paulo Roberto Garcia Lucareli, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PL001
Record Dates: First submitted 2013-02-28; First posted 2013-03-05 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sensorimotor (Experimental): Sensorimotor, this arm will receive sensorimotor and hip muscle strengthening.
  Interventions: Other: Sensorimotor
- Strength (Active Comparator): Strength, this arm will receive only hip muscle strengthening.
  Interventions: Other: Strength

INTERVENTIONS:
Other: Strength
  Other Names: Hip abductors and lateral rotators and knee extensors strengthening
  Arms: Strength
Other: Sensorimotor
  Other Names: Sensorimotor, balancing exercises, motor coordination, proprioceptive stimuli.
  Arms: Sensorimotor

SUMMARY:
Assess pain, function, trunk and lower limbs kinematic during functional tasks after hip muscle strengthening versus hip muscle strengthening and sensory motor training in lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary women,
* previous knee pain last 3 months in at least two of the following activities: sitting for long periods, walk up or down stairs, squat, running and jumping

Exclusion Criteria:

* Lower limb surgery,
* patella displacement
* knee instability
* Heart or locomotor disorders which might influence the evaluation

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Function and pain intensity | 4 weeks

SECONDARY OUTCOMES:
Muscle strength of the hip and knee muscles | 4 weeks
Three-dimensional kinematics of the trunk and lower limbs during the step down task | 4 weeks
Function and pain intensity | 3 and 6 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Rabelo ND, Lima B, Reis AC, Bley AS, Yi LC, Fukuda TY, Costa LO, Lucareli PR. Neuromuscular training and muscle strengthening in patients with patellofemoral pain syndrome: a protocol of randomized controlled trial. BMC Musculoskelet Disord. 2014 May 16;15:157. doi: 10.1186/1471-2474-15-157. PMID 24884455
- See also: Related Info — http://www.uninove.br